CLINICAL TRIAL: NCT04521192
Title: A Bridging Study on the Bioequivalence of Fluzoparib Capsules With Different Specifications in Healthy Volunteers
Brief Title: Bioequivalence of Fluzoparib(SHR3162) Study on Healthy Chinese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FZPL-I-BE-001
Record Dates: First submitted 2020-08-19; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — fluzoparib

STUDY DESIGN:
Intervention Model Description: Single dose of oral administration of fluzoparib capsules
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR sequence group (Experimental)
  Interventions: Drug: Fluzoparib
- RT sequence group (Experimental)
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Fluzoparib — the first period: test preparation; the second period: reference preparation
  Arms: TR sequence group
Drug: Fluzoparib — the first period: reference preparation the second period: test preparation
  Arms: RT sequence group

SUMMARY:
The primary objective of the study is to evaluate the bioequivalence of two different specification of reference preparation capsules (10 mg/capsule, 40 mg/capsule and 100 mg/capsule, 1 capsule each) and test preparations capsules (50 mg/capsule×3). Two different specifications of fluzoparib was provided by Jiangsu HengRui Pharmaceutical Co., Ltd.

The secondary objective of the study is to evaluate the safety of test preparations and reference preparation fluzoparib capsules of different specifications in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the study, and fully understand the study content, process and possible adverse reactions;
2. Able to complete the research in accordance with the requirements of the study protocol;
3. Healthy male or female subjects aged 18-50 (including 18 or 50 years old) at the date of signing the informed consent;
4. The subject is willing to have no pregnancy plan in the next 6 months and voluntarily take effective contraceptive measures
5. Body weight ≥ 45kg, body mass index (BMI) within the range of 18 ~ 28kg /m2 (including 18 and 28);
6. Health status: no history of heart, liver, kidney, digestive tract, nervous system, mental disorders, and metabolic disorders;
7. No abnormalities in physical examination or abnormalities without clinical significance;
8. Creatinine clearance rate (CLCr) ≥70 mL/min;
9. Negative pregnancy test for women of child-bearing age;

Exclusion Criteria:

1. Pregnant and lactating women, women who have unprotected sex in the 14 days before screening;
2. Participated in blood donation within 3 months before screening and donated blood volume ≥400mL or blood loss ≥400mL, or received blood transfusion;
3. Allergies, including those with a history of severe drug allergy or drug allergy; a history of allergy to fluzoparib capsules or its excipients.
4. Have a history of drug and/or alcohol abuse; alcoholics (drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of liquor, or 100 mL of wine; smoking ≥ 5 cigarettes per day) or Those who cannot ban smoking and alcohol during the trial;
5. Those who have a history of cardiovascular diseases such as myocarditis, coronary heart disease, pathological arrhythmia, and stroke;
6. Lung diseases, including invasive lung disease, pneumonia, dyspnea, etc;
7. History of chronic kidney disease, renal impairment, and renal anemia;
8. There is a history of dysphagia or any gastrointestinal disease that affects drug absorption;
9. Any uncontrolled peptic ulcer, colitis, pancreatitis, etc;
10. Those who have undergone any surgery within 6 months before screening;
11. A clear medical history of other important organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system (such as uncontrolled diabetes, high blood pressure, etc.), so that the investigator Those who think it is not suitable to participate in this research;
12. Hepatotoxic drugs (such as dapsone, erythromycin, fluconazole, ketoconazole, rifampin) taken within 6 months before screening;
13. Those who have taken any clinical trial drugs within 3 months;
14. Any drug that changes liver enzyme activity was taken 28 days before or during the study period;
15. Take any prescription or over-the-counter drugs 7 days before taking the study drug;
16. Ingested any vitamin products or herbs 7 days before taking the study drug
17. Clinical laboratory tests are abnormal and clinically significant, or other clinical findings show the following diseases (including but not limited to gastrointestinal, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular disease);
18. Combined with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive) or combined with syphilis infection
19. Drinking grapefruit juice and beverages containing xanthine, caffeine, and alcohol 48 hours before taking the study drug, exercising vigorously, or having other factors affecting drug absorption, distribution, metabolism, and excretion;
20. The investigator believes that there are other factors that not suitable for participating in this trial;
21. Screening for alcohol and drug use was positive or had a history of drug abuse in the past five years or had used drugs in the 3 months prior to the trial;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Fluzoparib | Up to Day 10
Area Under the Plasma Concentration(AUC) of Fluzoparib | Up to Day 10

SECONDARY OUTCOMES:
Adverse events | Up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated hospital of QingDao university, Qingdao, Qingdao, China